CLINICAL TRIAL: NCT03064061
Title: Impact of a Virtual Reality Experience, Before Oocytes Retrieval for In-vitro Fertilisation Treatment, on Anxiety and on the Pregnancy Rate
Brief Title: Impact of Virtual Reality Before Oocytes Retrieval on Anxiety and Pregnancy Rate
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Principal Investigator, Roelants, MD, Cliniques universitaires Saint-Luc- Université Catholique de Louvain
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2016/20JUL/346
Record Dates: First submitted 2016-12-26; First posted 2017-02-24 (Actual); Last update posted 2018-03-22 (Actual); Status verified 2018-03

CONDITIONS: Anxiety; in Vitro Fertilization; Virtual Reality
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Reality Neutral (Sham Comparator): neutral VR session before oocytes retrieval
  Interventions: Device: Virtual reality
- Virtual reality Anxiety (Active Comparator): VR session with the goal of reducing anxiety before oocytes retrieval
  Interventions: Device: Virtual reality

INTERVENTIONS:
Device: Virtual reality — a device with virtual reality is given to the patients with a film of 18 minutes

SUMMARY:
The primary objective of this study is to evaluate the impact of a session of virtual reality (VR) with the objective of lowering the anxiety level on the clinical pregnancy rate following an In-vitro fertilisation (IVF) procedure. Indeed, anxiety in relation to infertility happens frequently and over time, can become stressful for our patients. This level of stress influences the effect of the infertility treatment. Reducing anxiety levels could promote the ability of the patients to face this stress and promote a greater chance of pregnancy in that context.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients benefiting from an oocytes retrieval as part of their IVF at Cliniques universitaires Saint-Luc.
* Simple IVF / IVF Intracytoplasmic sperm injection (ICSI)

Exclusion Criteria:

* Patients with long-term psychotherapeutic treatment
* Patients taking psychotropic drugs
* patient blind and deaf

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 600 (Estimated)
Dates: Start 2017-02-17 (Actual); Primary Completion 2019-03 (Estimated); Study Completion 2019-06-30 (Estimated)

PRIMARY OUTCOMES:
impact of the virtual reality on the pregnancy rate (Ultrasound) | 12 weeks
  measured by ultrasound

SECONDARY OUTCOMES:
impact of the virtual reality on anxiety (numeric scale) | immediate
  measured with numeric scale (0-10) before and after the VR
impact of the virtual reality on satisfaction | immediate
  measured by a numeric scale 0-10
impact of the virtual reality on pregnancy test | 6 weeks
  measured by blood beta HCG level
state-trait Anxiety Inventory | immediate
  measured with STAI Y-A Spielberger before and after the VR and when leaving the hospital

CONTACTS AND LOCATIONS:
Locations (1):
- Cliniques universitaires Saint-luc, Brussels, Belgium